CLINICAL TRIAL: NCT06589557
Title: Modern Diagnostic Methods and Evaluation of Rehabilitation Effects Using Virtual Reality (VR) Therapy for Patients With Cervical Spine Discopathy
Brief Title: Diagnostic Methods and VR Therapy for Cervical Spine Discopathy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Andżelina Wolan-Nieroda, Principal Investigator, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uniwersytet Rzeszowski
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Disability Evaluation; Recovery of Function
Keywords: Cervical Spine Discopathy; Virtual Reality Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: VR Therapy and Standard Rehabilitation (Other): Standard Rehabilitation supplemented with VR Therapy
  Interventions: Other: Virtual Reality (VR) and Standard Rehabilitation; Other: Standard Rehabilitation
- Control: Standard Rehabilitation (Other): Control group - Standard Rehabilitation, without VR Therapy
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Other: Virtual Reality (VR) and Standard Rehabilitation — VR Rehabilitation:
  The VR therapy includes exercises designed to improve the range of motion, coordination, and spatial awareness of the cervical spine. Each patient will complete 15 training sessions over three weeks (5 sessions per week, 2 hours per session), with an additional 30 minutes of daily VR exercises.
  Standard Rehabilitation Program:
  Manual Therapy: Mobilization and manipulation techniques are applied to enhance the mobility of the cervical spine joints.
  Proprioceptive Exercises: These exercises focus on improving body position awareness, movement, and balance.
  Strengthening and Stretching Exercises: Individually tailored exercises are provided to strengthen and stretch the neck muscles.
  Arms: Experimental: VR Therapy and Standard Rehabilitation
Other: Standard Rehabilitation — Patients in this group will participate solely in the standard rehabilitation program.
  Standard Rehabilitation Program:
  Number of Sessions: Each patient will complete 15 training sessions, held 5 times per week for 3 weeks, with each session lasting 2 hours.
  Program Components:
  Manual Therapy: Mobilization and manipulation techniques will be applied to improve the mobility of the cervical spine joints.
  Proprioceptive Exercises: These exercises aim to enhance body position awareness, movement control, and balance.
  Strengthening and Stretching Exercises: Customized exercises will be provided to strengthen and stretch the neck muscles, tailored to individual needs.

SUMMARY:
The study will assess modern diagnostic methods and evaluate the rehabilitation effects of virtual reality (VR) therapy in patients with cervical spine discopathy.

DETAILED DESCRIPTION:
Study Design and Group Composition:

The study will involve 100 patients with cervical spine discopathy participating in a rehabilitation program at the Provincial Hospital in Tarnów, Poland.

Eligible patients will be randomly assigned to one of two groups:

Study Group (50 patients): Participants will undergo a standard rehabilitation program supplemented with additional VR therapy aimed at improving the range of motion of the cervical spine.

Control Group (50 patients): Participants will only partake in the standard rehabilitation program.

Therapeutic Program:

Number of Therapy Sessions: Each patient will participate in a program consisting of 15 sessions (5 sessions per week for 3 weeks), with each session lasting 2 hours.

Patients in both groups will engage in the following therapies:

Manual Therapy: Techniques of mobilization and manipulation to enhance joint mobility in the cervical spine.

Proprioceptive Exercises: Exercises aimed at improving body position awareness, movement, and balance.

Individually Tailored Strengthening and Stretching Exercises: Focused on strengthening and stretching the neck muscles.

In addition, patients in the study group will participate in VR training:

VR Training: Exercises in a virtual environment designed to improve range of motion, coordination, and spatial awareness. Each VR session will last 30 minutes. Differences in outcomes between the two groups will allow for evaluating the additional impact of VR on improving cervical spine function.

Assessment Procedures:

Assessments will be conducted twice: before the therapy begins and after the rehabilitation program ends. Patients will undergo the following evaluations:

Diagnostic Measurements:

Goniometer CROM (Cervical Range of Motion): A specialized diagnostic device used for precise assessment of cervical spine range of motion in three planes: sagittal (flexion and extension), horizontal (left and right rotation), and frontal (left and right lateral bending). It uses a head attachment and magnetic collar to measure angles with 1° accuracy, crucial for precise diagnosis and treatment planning.

Zebris Device: A modern diagnostic tool combining marker technology and ultrasonic signals to comprehensively assess cervical spine mobility in all planes. Special markers on the patient's head are tracked by sensors, and the software processes this data to provide detailed information on movement ranges and directions.

VR Goggles: Used to assess cervical spine range of motion, vision, and proprioception. They create an interactive virtual environment, allowing for precise movement analysis and providing real-time feedback to the patient.

Functional Assessment Questionnaires:

Personal Data Survey: Collects basic information such as age, gender, medical history, current treatment, lifestyle, and other factors that may affect therapy.

VAS Pain Scale (Visual Analogue Scale): A tool for self-assessment of pain, where patients indicate their pain level on a line from 0 (no pain) to 10 (worst possible pain).

Neck Disability Index (NDI): Assesses the degree of disability and functional limitations through ten questions related to daily life activities.

SF-20 Quality of Life Scale: Evaluates general health and quality of life across six dimensions: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, mental health, and general health perceptions.

Study Procedure:

Diagnostic Evaluation:

Assessment of the repeatability and accuracy of diagnostic devices on healthy volunteers (100) and patients with cervical spine discopathy (100), using:

Goniometer CROM for precise measurement of cervical spine range of motion. Zebris device using marker systems and ultrasonic signals to assess mobility in all cervical spine planes.

VR goggles to evaluate cervical spine range of motion, vision, and proprioception.

Patient Information: Before testing, patients will be informed about the study's purpose and procedures, including the use of Goniometer CROM, Zebris device, and VR goggles.

Patient Positioning: Assessments will be conducted in a seated position with back support, feet flat on the floor, and hands resting on thighs to maintain a stable and comfortable posture.

Test Procedure:

Cervical Spine Mobility Assessment: Using the Goniometer CROM, Zebris device, and VR goggles to measure cervical spine movement in all planes (flexion, extension, left-right rotation, and left-right lateral bending).

Vision Range Assessment: Using VR goggles, patients will track moving objects across different parts of their visual field.

Proprioception Assessment with VR Goggles: Patients will replicate movements previously measured during the test to evaluate their depth perception and spatial coordinatio

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 65 years.
* Diagnosed and confirmed cervical spine discopathy (ICD-10: M50) through imaging studies (X-ray, MRI).
* Presence of symptoms related to cervical spine dysfunction, such as neck pain, limited range of motion, and radiating pain to the arms.
* Informed consent to participate in the study and willingness to adhere to rehabilitation recommendations.

Exclusion Criteria:

* Active rheumatic diseases, cancers, advanced diabetes, cardiovascular diseases, or other conditions affecting the safety and effectiveness of rehabilitation.
* Cervical spine surgeries performed within the last 6 months.
* Cervical spine injuries, including fractures or dislocations.
* Severe mental disorders.
* Lack of informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of cervical spine range of motion using a Cervical Range of Motion (CROM) goniometer and the Zebris system. | First examination - before the start of the rehabilitation program;
  Assessment of cervical spine mobility in all planes (flexion, extension, lateral bending, and rotation).
  Unit of Measure: Range of motion measured in degrees (°), indicating the exact angles of neck movement in each direction.
  Measurement Tool: The Cervical Range of Motion (CROM) goniometer and Zebris device will be used to measure the exact angles of neck movement with an accuracy of 1°. These tools will evaluate cervical spine mobility across all planes of movement.
Assessment of cervical spine range of motion using a Cervical Range of Motion (CROM) goniometer and the Zebris system. | Second examination - at the end of the three-week program
  Assessment of cervical spine mobility in all planes (flexion, extension, lateral bending, and rotation).
  Unit of Measure: Range of motion measured in degrees (°), indicating the exact angles of neck movement in each direction.
  Measurement Tool: The Cervical Range of Motion (CROM) goniometer and Zebris device will be used to measure the exact angles of neck movement with an accuracy of 1°. These tools will evaluate cervical spine mobility across all planes of movement.
Assessment of cervical spine proprioception using virtual reality (VR) goggles. | First examination - before the start of the rehabilitation program;
  Assessment of deep neck sensation and the ability to perceive the position and movement of the neck. Unit of Measure: Deviation from the intended neck movement measured in degrees (°), which the patient can replicate during proprioceptive tests.Measurement Tool: Virtual Reality (VR) goggles will be the sole tool used to conduct proprioceptive tests. Patients will replicate neck movements displayed in the virtual environment, and the accuracy of these movements will be measured in degrees to assess proprioception and spatial coordination.
  Method: Using VR goggles to conduct proprioceptive tests, where patients replicate movements shown in the virtual environment to assess their depth perception and spatial coordination.
Assessment of cervical spine proprioception using virtual reality (VR) goggles. | Second examination - at the end of the three-week program
  Assessment of deep neck sensation and the ability to perceive the position and movement of the neck. Unit of Measure: Deviation from the intended neck movement measured in degrees (°), which the patient can replicate during proprioceptive tests.Measurement Tool: Virtual Reality (VR) goggles will be the sole tool used to conduct proprioceptive tests. Patients will replicate neck movements displayed in the virtual environment, and the accuracy of these movements will be measured in degrees to assess proprioception and spatial coordination.
  Method: Using VR goggles to conduct proprioceptive tests, where patients replicate movements shown in the virtual environment to assess their depth perception and spatial coordination.
Assessment of visual field during neck movements using virtual reality (VR) goggles. | First examination - before the start of the rehabilitation program;
  Measurement of the range of vision while performing neck movements, with the patient seated and looking straight ahead.
  Unit of Measure: Range of vision measured in degrees (°), indicating the extent to which the patient can perceive moving objects in different parts of their visual field while maintaining a forward gaze.
  Measurement Tool: Virtual Reality (VR) goggles will be used to track and analyze the patient's ability to follow moving objects across their visual field while sitting and looking straight ahead. The visual range will be measured in degrees to assess the field of vision during neck movements without changing the direction of the gaze.
Assessment of visual field during neck movements using virtual reality (VR) goggles. | Second examination - at the end of the three-week program
  Measurement of the range of vision while performing neck movements, with the patient seated and looking straight ahead.
  Unit of Measure: Range of vision measured in degrees (°), indicating the extent to which the patient can perceive moving objects in different parts of their visual field while maintaining a forward gaze.
  Measurement Tool: Virtual Reality (VR) goggles will be used to track and analyze the patient's ability to follow moving objects across their visual field while sitting and looking straight ahead. The visual range will be measured in degrees to assess the field of vision during neck movements without changing the direction of the gaze

SECONDARY OUTCOMES:
Assessment of pain symptoms in the cervical spine region using the Visual Analog Scale (VAS). | First examination - before the start of the rehabilitation program;
  Evaluation of pain levels in the cervical spine region. Unit of Measure: Pain intensity is measured on a scale of 0 to 10 using the Visual Analogue Scale (VAS), where 0 represents no pain and 10 represents the worst pain imaginable.
  Measurement Tool: The Visual Analogue Scale (VAS) will be used to allow patients to self-report their perceived pain intensity in the cervical spine region
Assessment of pain symptoms in the cervical spine region using the Visual Analog Scale (VAS). | Second examination - at the end of the three-week program
  Evaluation of pain levels in the cervical spine region. Unit of Measure: Pain intensity is measured on a scale of 0 to 10 using the Visual Analogue Scale (VAS), where 0 represents no pain and 10 represents the worst pain imaginable.
  Measurement Tool: The Visual Analogue Scale (VAS) will be used to allow patients to self-report their perceived pain intensity in the cervical spine region
Assessment of functional improvement in daily activities and overall functionality using the Neck Disability Index (NDI) questionnaire. | First examination - before the start of the rehabilitation program;
  Assessment of the impact of therapy on daily activities and functionality related to neck pain.
  Unit of Measure: Functional limitations and disability levels are measured as a percentage (%) using the Neck Disability Index (NDI), where higher percentages indicate greater disability.
  Measurement Tool: The NDI assesses disability and functional limitations caused by neck pain, with 10 items scored from 0 to 5, for a maximum score of 50. The score is expressed as a percentage, with higher percentages indicating more severe disability:
  0-4 points (0-8%): No disability 5-14 points (10-28%): Mild disability 15-24 points (30-48%): Moderate disability 25-34 points (50-68%): Severe disability 35-50 points (70-100%): Complete disability.
Assessment of functional improvement in daily activities and overall functionality using the Neck Disability Index (NDI) questionnaire. | Second examination - at the end of the three-week program
  Assessment of the impact of therapy on daily activities and functionality related to neck pain.
  Unit of Measure: Functional limitations and disability levels are measured as a percentage (%) using the Neck Disability Index (NDI), where higher percentages indicate greater disability.
  Measurement Tool: The NDI assesses disability and functional limitations caused by neck pain, with 10 items scored from 0 to 5, for a maximum score of 50. The score is expressed as a percentage, with higher percentages indicating more severe disability:
  0-4 points (0-8%): No disability 5-14 points (10-28%): Mild disability 15-24 points (30-48%): Moderate disability 25-34 points (50-68%): Severe disability 35-50 points (70-100%): Complete disability.
Quality of life assessment using the SF-20 Health Survey questionnaire. | First examination - before the start of the rehabilitation program;
  Evaluation of general health and quality of life will be conducted across six dimensions: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, mental health, and general health perceptions.
  Unit of Measure: Scores for each dimension range from 0 to 100, with higher scores indicating better functioning and quality of life.
  Measurement Tool: The SF-20 Health Survey will be used to assess general health and quality of life. Each dimension is scored separately, with 0 indicating the poorest health or most severe limitations, and 100 representing the best health or no limitations. The score for each dimension is the average of the relevant questions, providing a detailed profile of the individual's health across each dimension, without a total combined score.
Quality of life assessment using the SF-20 Health Survey questionnaire. | Second examination - at the end of the three-week program
  Evaluation of general health and quality of life will be conducted across six dimensions: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, mental health, and general health perceptions.
  Unit of Measure: Scores for each dimension range from 0 to 100, with higher scores indicating better functioning and quality of life.
  Measurement Tool: The SF-20 Health Survey will be used to assess general health and quality of life. Each dimension is scored separately, with 0 indicating the poorest health or most severe limitations, and 100 representing the best health or no limitations. The score for each dimension is the average of the relevant questions, providing a detailed profile of the individual's health across each dimension, without a total combined score.

CONTACTS AND LOCATIONS:
Overall Officials: Andżelina Wolan-Nieroda, PhD, Principal Investigator — University of Rzeszow; Agnieszka Guzik, Professor, Study Chair — University of Rzeszow
Locations (1):
- Andżelina Wolan-Nieroda, Rzeszów, Al. Rejtana 16C, Poland

IPD SHARING:
Plan to Share IPD: No